CLINICAL TRIAL: NCT04731389
Title: Digital Strategies for Patients With Chronic Dermatosis With Pruritus / Skin Picking Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Carolina Blaya Dreher, Professor, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37827820.6.0000.5327
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Skin-Picking; Acne; Dermatosis
Keywords: skin picking; cognitive-behavioral therapy; internet-based therapy; psychodermatosis; acne
MeSH Terms: conditions — Excoriation Disorder; Acne Vulgaris; Skin Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internet CBT (Experimental): Intervention with remote and self-applicable cognitive behavioral therapy, during 4 weeks.
  Interventions: Behavioral: internet-based cognitive-behavioral therapy
- Quality of life promotion (Active Comparator): Control intervention, during 4 weeks.
  Interventions: Behavioral: Quality of life improving intervention

INTERVENTIONS:
Behavioral: internet-based cognitive-behavioral therapy — Composed of 4 modules: the first module will address psychoeducation on dermatillomania, self-monitoring of symptoms and habit reversal techniques; the second module works with anxiety coping techniques (diaphragmatic breathing and muscle relaxation); module 3 addresses cognitive correction techniques, such as stopping thinking, analyzing evidence, reassigning severity and responsibilities; the last module reviews the techniques learned and addresses techniques for preventing symptom relapse. The modules will be applied by the patient in an online format, each module lasts an average of 30 minutes. The platform will send notice by email through automation tools, SMS or message by application to patients to remind them to complete 1 module per week.
  Other Names: Active intervention group
  Arms: internet CBT
Behavioral: Quality of life improving intervention — consisting of videos with guidance on quality of life, with a total of 4 videos of 2 minutes, each being made available in 1 week, consisting of: guidance on sleep hygiene; guidance on healthy eating; guidelines on the practice of physical activity and guidelines on the excessive use of social networks.
  Other Names: Active control group
  Arms: Quality of life promotion

SUMMARY:
Almost 35% of patients treated to dermatosis have some psychiatric disorder. The aim of this study is to evaluate the prevalence and severity of skin picking disorder and other dermatosis, and also test the efficacy of an online-delivered cognitive-behavioral therapy to improve skin picking disorder severity.

DETAILED DESCRIPTION:
The interface between dermatology and psychiatry represents a major challenge for the management of chronic itchy pathologies. Dermatology requires adherence to chronic treatments that must be incorporated as changes in habit. In addition, patients with chronic pruritic dermatoses often develop a scratching habit that often leads to the development of dermatillomania, requiring psychiatric intervention. In general, among the patients who seek the dermatologist, 33% complain of psychiatric symptoms. On the other hand, patients with psychiatric conditions have a higher prevalence of dermatoses when compared to the healthy population, with anxiety, depression and psychosis being situations that can induce or worsen dermatological conditions. Despite the important interface between dermatology and psychiatry, there is still a gap in the literature about the best way to diagnose and treat these patients affected by psychodermatosis, and also a lack of professionals' knowledge about this theme. One study addressed the quality of the treatments currently offered for skin picking, also known as dermatillomania, finding that only 53% of patients report having received the correct diagnosis of their pathology, and after the treatment offered, 54.7% of individuals reported that their clinical condition was unchanged or worse, and only 11% of patients reported feeling better with the treatment performed. When asked about the training of professionals, 85% of patients reported that the professional did not seem to have knowledge about his clinical condition.

The current world moment, in the face of the Covid-19 pandemic, keeps these patients away from possible interventions that could bring relief to the situation, either for fear of contamination, difficulties in displacement or even a temporary reduction in vacancies for care. The great and just effort of the Health Systems to face the pandemic can, on the other hand, impact the offer of assistance to chronic dermatological diseases. Around the world, telemedicine and other distance health care protocols have been used in an attempt to assist patients. But not all carriers of these chronic diseases are part of health systems. It is also known that during the COVID pandemic19, dermatoses frequently associated with dermatillomania are still the most common causes of consultations with dermatologists, such as acne and eczema. Changes in routine, especially food and physical activity, but also in certain habits, such as frequent hand hygiene and the use of astringent substances, such as alcohol gel, worsen or trigger inflammatory conditions. Still, the frequent use of masks induces the appearance of pruritus, which can increase the severity of already existing dermatoses and, also, lead to the misuse of props.

Thus, the investigators propose the development of an electronic website with educational strategies and self-applicable tools for cognitive behavioral therapy to patients with dermatoses who have pruritus or symptoms on the skin with the potential to develop or even with the diagnosis of skin picking. The website proposed here aims to help patients with chronic dermatoses seeking both the prevention and treatment of possible complications. This set of Internet pages aims to provide educational material, strategies to increase adherence to treatment and interventions with cognitive-behavioral therapy techniques, facilitating patients' autonomy in caring for their skin disorders, especially in times as troubled as the current one.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years
* Internet access
* Diagnosis of Skin Picking (dermatillomania)
* Patients may be diagnosed or not with primary dermatoses, such as acne, atopic dermatitis, psoriasis and rosacea

Exclusion Criteria:

* Dementias
* Acute psychotic disorder, bipolar disorder in acute episode, psychoactive substance use disorder (except tobacco), severe depressive episode or suicidal ideation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Skin Picking Scale Revised | 6 months and 12 months
  Improvement in the severity of dermatillomania assessed by the Skin Picking Scale Revised, adapted to the Brazilian population.The scale scores vary from 0-32, with higher scores meaning more severe symptoms.

SECONDARY OUTCOMES:
Change in patient health questionnaire (PHQ-9) | 6 months and 12 months
  Improvement in depression assessed by the PHQ-9 scale. The scale scores vary from 0-27, with higher scores meaning more severe symptoms.
Change in General Anxiety Disorder-7 (GAD-7) | 6 months and 12 months
  Improvement in anxiety assessed by the GAD-7 scale. The scale scores vary from 0-21, with higher scores meaning more severe symptoms.
Change in Dermatology Life Quality Index (DLQI) | 6 months and 12 months
  Improvement in quality of life related to skin assessed by DLQI scale. The scale scoring vary from 0-30, with higher scoring meaning more severe life impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided